CLINICAL TRIAL: NCT05340556
Title: Microchimerism From a Firstborn Boy or an Older Brother in Patients With Recurrent Pregnancy Losses: a Pilot Study
Brief Title: Microchimerism in Patients With Recurrent Pregnancy Losses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Caroline Nørgaard-Pedersen (Other)
Collaborators: Department of Clinical Immunology, Odense University Hospital, DK (Unknown); Aalborg University Hospital (Other)
Responsible Party: Sponsor-Investigator, Caroline Nørgaard-Pedersen, Principal investigator, Aalborg University Hospital
Organization: Aalborg University Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: F2022-012
Record Dates: First submitted 2022-04-08; First posted 2022-04-22 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-10

CONDITIONS: Recurrent Pregnancy Loss, Not Pregnant
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sRPL patient (Experimental): sRPL with an older brother and at least one child prior to diagnosis
  Interventions: Genetic: Blood sample
- Brother or child to the sRPL patient (Experimental): An older brother (with at least same biological mother) og child to the sRPL patient
  Interventions: Genetic: Swap test

INTERVENTIONS:
Genetic: Blood sample — Blood sample of 12 ml EDTA plasma.
  Arms: sRPL patient
Genetic: Swap test — receive swab tests for collecting cells from the oral mucosa
  Arms: Brother or child to the sRPL patient

SUMMARY:
This pilot study aims to evaluate if microchimeric cells in a patient with recurrent pregnancy loss (RPL) can be detected by the blood analysis for the presence of the DYS14 gene and the use of indel-panel methods and also, to examine if this method can distinguish the cell's origin; comparing gene sequence from the patient's firstborn son or her older brother. In addition, the pilot study will provide the investigators with information and experience necessary for a subsequent main study to be conducted.

DETAILED DESCRIPTION:
To the investigators' knowledge, no previous study has determined the origin of microchimeric cells, and therefore, this pilot study will use a newly developed genetic analysis which will compare DNA fragments from the male microchimeric cells with DNA fragments from the RPL patient's son(s) and older brother(s).

The pilot study aims to evaluate the functions and capacity of a newly developed genetic test identifying microchimeric cells. A pilot study is necessary to assure the DNA fragments (indels) analyzed in the genetic analysis include enough informative differences to distinguish between the son(s), daughter(s) and the older brother(s) before these investigations can be initiated in a larger sample. To assure the test can distinguish origin of microchimeric cells between relatives and work independent of gender, The study will include both the proband's daughter(s) and son(s) to strengthen the confidence that the test possesses this ability.

10 sRPL and their older brother(s) and firstborn child is included. total included: approx 30.

Only sRPL whose brother(s) and child(ren) also consent to participate, will be included.

Blood sample of 12 ml EDTA plasma is collected from the sRPL patient. A swap sample from oral mucosa is collected from the older brother and child(ren).

The samples will be centrifuged and the buffy coat containing the DNA will be collected from patient and stored at -80 °C. To detect the multi-copy DYS14 marker located in the TSPY1 gene on the Y-chromosome a real-time PCR analysis will be performed on the extracted DNA with a PCR mastermix specific for the reference gene.

Also, The extracted DNA will be amplified using specific primers and their associated probes in a multiplex PCR analysis. The specific primers target the 10 different indels leading to 10 PCR products with non-overlapping amplicon sizes. After the PCR analyses, the fragments are analyzed by capillary electrophoresis using GeneticAnalyzer and GeneMapper. When differences are identified, a qPCR analysis is performed on samples from only the proband with primers and probes specific for the indel fragments that are only present in either the child or the older brother. 12 wells loaded with 30.000 GE in each well are screened along with a no-template control and a positive control containing 10 GE of DNA homozygous for the allele variant.

ELIGIBILITY:
sRPL patient (proband):

Inclusion Criteria:

* ≥3 consecutive pregnancy losses ≤12 weeks of gestation, which do not include confirmed ectopic or molar pregnancies.
* Age <41 years at time of admission
* Patients who have minimum one alive older brother with a common mother and prior birth of a boy, and patients who have minimum one alive older brother with a common mother and prior birth of a girl.

Exclusion Criteria:

* Significant intrauterine malformations
* Thyroid dysfunction
* Known chromosomal abnormality
* An older brother, a son or a daughter from whom we cannot not collect a swab test e.g., due to lack of consent, death, distance etc.
* Transplant recipient
* Transfusion recipient
* Pregnancy at the time the blood sample is collected

Older Brother:

Inclusion Criteria:

* Age difference between proband and the older brother <15 years
* Common mother with the proband

sRPL patient's child:

Inclusion Criteria:

* Age <15 years

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — sRPL patient: women. Sibling: Older brother to sRPL patient. Child: The sRPL patient's child(ren) of both sexes. Biological sex is used.
Enrollment: 32 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2024-02-05 (Actual); Study Completion 2024-02-05 (Actual)

PRIMARY OUTCOMES:
Frequency of sRPL patients with microchimeric male cells | Non-pregnant state, performed during study completion, i.e. within 1 year
  Prevalence of sRPL patients with microchimeric male cells in the peripheral blood
Frequency of sRPL patients with microchimeric cell originating from older brother | Non-pregnant state, performed during study completion, i.e. within 1 year
  Determination of microchimeric cell origin: brother, son, daughter or not identified
Frequency of sRPL patients with microchimeric cell originating from the patient's son | Non-pregnant state, performed during study completion, i.e. within 1 year
  Determination of microchimeric cell origin: brother, son, daughter or not identified
Frequency of sRPL patients with microchimeric cell originating from the patient's daughter | Non-pregnant state, performed during study completion, i.e. within 1 year
  Determination of microchimeric cell origin: brother, son, daughter or not identified
Frequency of sRPL patients with microchimeric cell originating from unknown person | Non-pregnant state, performed during study completion, i.e. within 1 year
  Determination of microchimeric cell origin: brother, son, daughter or not identified

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Nørgaard-Pedersen, MD, Principal Investigator — Aalborg University Hospital, Denmark
Locations (1):
- Aalborg University Hospital, Aalborg, Denmark